CLINICAL TRIAL: NCT06834438
Title: An Open- Label, Single-arm, Dose-escalation Pilot Study to Evaluate the Safety, Tolerability and Preliminary Efficacy of ST002 in the Treatment of Patients with NF2 Mutation-related Solid Tumors
Brief Title: Gene Therapy for Neurofibromatosis Type 2 (NF2) with ST002
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, NING LI, Vice president of Cancer Hospital Chinese Academy of Medical Sciences, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ST002-IIT-2024-01
Record Dates: First submitted 2025-02-07; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: NF2 Deficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- ST002 (Experimental): Subjects will receive with a single multi-point intra-tumoral injection of ST002 from 1x10^7 to 1x10^8 TU into the tumor.
  Interventions: Genetic: ST002

INTERVENTIONS:
Genetic: ST002 — Single multi-point intra-tumoral injection of ST002, a lentiviral vector designed to drive expression of the NF2 protein product, Merlin.

SUMMARY:
This is an open-label, single-arm, dose-escalation pilot study to evaluate the safety, tolerability and preliminary efficacy of ST002 in the treatment of patients with NF2 mutation-related solid tumors. ST002 injection is a gene therapy product designed for NF2. By reinserting the normal XXX gene into genetically deficient tumor cells, the product expresses Merlin. This regulates gene transcription in tumor cells, controls the tumor microenvironment, and inhibits tumor growth and invasion, achieving therapeutic effects.

DETAILED DESCRIPTION:
This is an open-label, single-arm, dose-escalation pilot study to evaluate the safety, tolerability and preliminary efficacy of ST002 in the treatment of patients with NF2 mutation-related solid tumors. Using a 3+3 dose escalation design, three dose groups are formulated, and three to six patients are expected to be enrolled in each dose group. A total of nine to eighteen - patients with NF2 gene mutation related solid tumors will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* age ≥16 years old, gender not limited;
* Patients must meet the diagnostic criteria for NF2 gene mutations, which are benign or malignant solid tumors with confirmed NF2 gene mutations or no expression of the NF2 protein product Merlin in peripheral blood or tumor tissue, and no standard treatment or with standard treatment failure;
* at least one measurable and injectable superficial lesion (according to RECIST or itRECIST criteria);
* Having sufficient organ and bone marrow function:

  1. Blood routine (no transfusion or treatment with colony-stimulating factor within 14 days): neutrophil count (ANC) ≥ 1.5 × 10 9 /L, hemoglobin (Hb) ≥ 90g/L, platelet count (PLT) ≥ 75 × 10 9 /L; White blood cell count (WBC)>3.0 × 10 9 /L;
  2. Liver function: Serum total bilirubin (TBIL) ≤ 1.5 × ULN, ALT≤2.5×ULN， AST ≤ 2.5 × ULN (ALT ≤ 5 × ULN, AST ≤ 5 × ULN in patients with liver metastasis);
  3. Renal function: serum creatinine (Cr) ≤ 1.5 × ULN, or creatinine clearance rate (CrCl) ≥ 50ml/min; d) Coagulation function: Prothrombin time (PT) ≤ 1.5 × ULN, activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, international normalized ratio (INR) ≤ 1.5 × ULN;
* Patients must voluntarily participate in clinical trials, demonstrate adherence to the study protocol, cooperate well with researchers, and sign a written informed consent form.

Exclusion Criteria:

* Has participated in or is currently participating in other clinical studies NF2 targeting gene therapy;
* History of severe neurological disorders such as epilepsy (excluding neurofibromatosis);
* Patients who are allergic to lentiviral vectors and their excipients;
* Patients with poorly controlled hypertension (systolic blood pressure>150 mmHg and/or diastolic blood pressure>100 mmHg under regular medication control), as well as those with a history of hypertensive crisis or hypertensive brain disease;
* Suffering from unstable angina or acute myocardial infarction, or having a history of both within the past six months;
* Patients with a history of malignant tumors within the past 5 years, except for cured basal cell carcinoma, squamous cell carcinoma of the skin, cervical cancer, and gastrointestinal cancer;
* During the study period, premenopausal women who are pregnant, breastfeeding, has a positive pregnancy test, or are unwilling to take contraceptive measures.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Safety evaluation | From baseline to Week 24 after administration
  Evaluate the incidence of drug-related adverse events (AEs) and adverse events (SAEs) from baseline to Week 24 after administration, with a focus on neurotoxicity and genome-wide integration carcinogenic risks.

SECONDARY OUTCOMES:
Efficacy evaluation | Day 21 after administration, and at the end of study follow-up, and at early withdrawal. The frequency of checks during the research period can be adjusted according to the researcher's judgement.
  Evaluate the objective response rate (ORR) (tumor volume reduction) and duration of response (DOR) according to RECIST and itRECIST
Efficacy evaluation | Day 21 after injection
  Percentage of necrosis of tumor cells in the tumor tissue at the injection site, estimated by pathological HE staining, at Day 21 after administration.

CONTACTS AND LOCATIONS:
Overall Officials: Shuhang Wang, PhD, Study Director — National Cancer Center of China
Locations (1):
- Shuhang Wang, Beijing, Beijing Municipality, China